CLINICAL TRIAL: NCT03464266
Title: Impact of Concurrent Initiation of DMPA Contraception and Tenofovir PrEP on Bone Loss in Young Women
Brief Title: The Kampala Women's Bone Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Makerere University (Other); MU-JHU CARE (Other); Columbia University (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Renee Heffron, Assistant Professor, Global Health and Epidemiology, University of Washington
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00001451; R01HD089843 (NIH)
Record Dates: First submitted 2018-02-25; First posted 2018-03-14 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Bone Demineralization; Hypoestrogenism; Subclinical Kidney Injury; Bone Microarchitecture
MeSH Terms: conditions — Bone Demineralization, Pathologic | interventions — N,N-dimethyl-4-anisidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- DMPA and PrEP (Active Comparator)
  Interventions: Combination Product: FTC/TDF and DMPA
- DMPA and no PrEP (Active Comparator)
  Interventions: Drug: DMPA
- Condoms only and PrEP (Active Comparator)
  Interventions: Drug: FTC/TDF
- Condoms only and no PrEP (Active Comparator)
  Interventions: Other: Neither DMPA nor FTC/TDF

INTERVENTIONS:
Combination Product: FTC/TDF and DMPA — The primary analysis will be separate comparisons of the annualized rates of change in BMD and TBS of the spine and hip between women using PrEP and DMPA concurrently versus women using DMPA only (comparison 1), women using PrEP only (comparison 2), and women using neither (comparison 3). Analyses will account for baseline BMD.
  Arms: DMPA and PrEP
Drug: FTC/TDF — The primary analysis will be separate comparisons of the annualized rates of change in BMD and TBS of the spine and hip between women using PrEP and DMPA concurrently versus women using DMPA only (comparison 1), women using PrEP only (comparison 2), and women using neither (comparison 3). Analyses will account for baseline BMD.
  Arms: Condoms only and PrEP
Drug: DMPA — The primary analysis will be separate comparisons of the annualized rates of change in BMD and TBS of the spine and hip between women using PrEP and DMPA concurrently versus women using DMPA only (comparison 1), women using PrEP only (comparison 2), and women using neither (comparison 3). Analyses will account for baseline BMD.
  Arms: DMPA and no PrEP
Other: Neither DMPA nor FTC/TDF — The primary analysis will be separate comparisons of the annualized rates of change in BMD and TBS of the spine and hip between women using PrEP and DMPA concurrently versus women using DMPA only (comparison 1), women using PrEP only (comparison 2), and women using neither (comparison 3). Analyses will account for baseline BMD.
  Arms: Condoms only and no PrEP

SUMMARY:
The primary objective of this study is to address critical safety questions with concurrent TDF-based PrEP and DMPA use. We hypothesize that young women using TDF-based PrEP and DMPA will have lower bone acquisition and altered bone metabolism. Bone mineral metabolism is in part regulated by the kidney, and we hypothesize that bone effects from concurrent PrEP and DMPA use will be driven by subclinical kidney injury, a known side effect of TDF, as well as DMPA-induced hypoestrogenism. To investigate our hypothesis, we will enroll a prospective cohort of approximately 500 HIV-uninfected women ages 16-25 years in Kampala, Uganda who have substantial HIV risk and are initiating DMPA or barrier method contraception. Over a 24-month period, we will offer TDF-based PrEP. We will use state-of-the-art radiologic, biochemical, and epidemiologic methods to test the hypothesis that concurrent TDF-based PrEP and DMPA use results in compounding adverse effects on bone health.

DETAILED DESCRIPTION:
The proposed research will investigate the hypothesis that TDF-based PrEP and DMPA initiated concurrently by HIV-uninfected women will enhance each other's effects on bone metabolism. The investigators will conduct an open-label prospective study of approximately 500 HIV-uninfected women at substantial risk for HIV-infection who are newly initiating DMPA or using condoms as their only contraceptive in Kampala, Uganda. The investigators will offer PrEP to all of these women and determine the joint effect of PrEP and DMPA on changes in bone mass (Aim 1), bone turnover, subclinical kidney injury, and hypoestrogenism (Aim 2), and conduct mediation analysis to assess the contribution of each pathway to overall losses in bone mass (Aim 3).

1. The investigators will assess whether young women using TDF-based PrEP and DMPA concurrently attain lower peak bone mass over a 24-month period and have evidence of disrupted microarchitecture, relative to women using either agent singly or neither agent The investigators will use dual energy x-ray absorptiometry (DXA) scans to measure BMD annually at 3 anatomical sites (lumbar spine, total hip, and wrist). Additionally, the investigators will derive the trabecular bone score (TBS), an index of lumbar spine trabecular microarchitecture.
2. The investigators will investigate whether young women concurrently using TDF-based PrEP and DMPA experience: 1) higher rates of bone turnover, a direct precursor to bone loss and 2) subclinical kidney injury and hypoestrogenism, markers of two mechanistic pathways between TDF and DMPA use and bone mass

At baseline and 24 months, the investigators will measure:

1. Markers of bone formation and resorption (e.g. NTX, P1NP, serum intact parathyroid hormone, total and bioavailable 25-OH-vitamin D)
2. Markers of kidney function (phosphate, glucose, creatinine, total protein, albumin) and
3. Markers of estrogen (serum estradiol, sex hormone binding protein, and the occurrence of amenorrhea) Hypothesis: Relative to women using DMPA only and PrEP only, women concurrently using TDF-based PrEP and DMPA will have increased bone turnover markers and PTH. In addition, women concurrently using TDF-based PrEP and DMPA will have more frequent subclinical kidney injury (relative to women without tenofovir exposure) and reduced serum estrogen (relative to women without DMPA exposure).

3. Using mediation analysis, the investigators will identify the degree to which the pathways through subclinical kidney injury and hypoestrogenism account for changes in bone density among women concurrently using TDF-based PrEP and DMPA The investigators will conduct mediation analysis to determine the degree to which changes in the pathways through subclinical kidney injury, hypoestrogenism and the combination of these pathways account for changes in bone density.

Over a 24-month period, the investigators will follow women quarterly with HIV rapid testing, PrEP adherence counseling and refills, DMPA injections, and provision of other contraceptives as desired. At enrollment and quarterly visits, the investigators will assess physical activity, sexual behavior, and menstrual cycle characteristics. Annually, the investigators will conduct physical exams and anthropometric readings. Sexually transmitted infections will be routinely assessed syndromically, according to national guidelines. Women will be encouraged to consider their HIV risk and fertility desires at every visit and counseled about contraception and PrEP accordingly. Dual energy x-ray absorptiometry (DXA) scans will be performed at baseline and annually thereafter. Blood and urine samples will be obtained quarterly, aliquoted, and archived at minus 80o Celsius.

DXA and TBS assessments:

DXA scans will be conducted at study enrollment (within 1 week of contraceptive initiation), 12, and 24 months after enrollment. DXA is the clinical standard for measuring BMD. It is painless and non-invasive. Women will be exposed to a relatively low level of radiation which is <1/10 the dose of a standard chest x-ray, and less than a day's exposure to natural radiation. BMD by DXA of the hip and spine is generally considered the most reliable way to classify osteoporosis, assess changes in BMD, and predict fracture risk. The investigators will measure areal BMD of the lumbar spine (L1-4), hip, and wrist, and body composition (total and % fat and lean mass) using a DXA machine. For the TBS analysis, no additional image acquisition is required. TBS will be performed as a re-analysis of the lumbar spine taken as part of the standard DXA procedure with specialized software.

Contraceptive provision:

Women will initiate contraception at the study clinic or a family planning clinic, as they are seeking services. Throughout study follow up, the study will assume responsibility for contraceptive provision, including DMPA injections, and care of all other methods desired by women. The staff at the IDI-Kasangati research clinic have extensive experience with the provision of contraception and contraceptive counseling during previous HIV prevention studies.

PrEP provision and adherence monitoring

Co-formulated emtricitabine FTC/TDF will be provided as PrEP by the study. PrEP counseling and provision will follow WHO guidelines, or Ugandan clinical guidelines when they are available. The investigators will measure adherence using three different methods:

1. Pill counts will be conducted by the pharmacist during study visits to determine the percentage of expected pills that were used
2. Real time monitoring will be conducted using an electronic monitoring system that captures a date-time stamp each time the pill container is opened
3. The primary circulating form of TDF, tenofovir (TFV), will be quantified in blood archives from 1) a random sample of up to 15% of women who initiate PrEP to characterize the adherence in the cohort overall and 2) a targeted group of women who have no BMD change and women who experience a fracture.

Laboratory processing to measure markers of bone turnover, subclinical kidney injury, and hypoestrogenism.

Using state-of-the-art assay techniques on archival samples, the investigators will measure 1) established markers of bone turnover and bone health, 2) markers of subclinical kidney injury, and 3) markers of hypoestrogenism. Archived samples will be batch-analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Age 16-25

If age 16-17:

* qualification as an emancipated minor (due to past pregnancy, being married, having a child, or catering for their own livelihood) or a mature minor (due to having a sexually transmitted infection) or able to have a parent/guardian provide informed consent
* HIV-uninfected
* Initiated DMPA within the past 90 days or using condoms only for contraception
* Willing and able to provide written informed consent
* Not planning to get pregnant in the next 24 months
* Sexually active
* Planning to remain in the study area for the next 2 years

Exclusion Criteria:

* Exclusion criteria:
* Currently enrolled in a biomedical HIV-1 prevention study
* Current or prior use of PrEP consecutively in the last 3 months
* Abnormal renal function (creatinine clearance <60 min/ml)
* Hepatitis B infection
* Currently pregnant or breastfeeding
* Current DMPA use for longer than 90 days
* Use of implant, IUD, or oral contraceptives
* Past hysterectomy, oophorectomy, or tubal ligation
* Current or recent history of primary or secondary amenorrhea
* Taking medications known to interfere with bone metabolism (steroids, anti-convulsants, bisphosphonates, cancer drugs).
* Has any other condition that would preclude the ability to provide informed consent, make study participation unsafe, complicate the interpretation of study findings or otherwise interfere with achievement of the study objectives, in the investigator's discretion.

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
The investigators will assess whether young women using TDF-based PrEP and DMPA concurrently attain lower peak bone mass over a 24-month relative to women using either agent singly or neither agent. | 24 months
  The investigators will use dual energy x-ray absorptiometry (DXA) scans to measure BMD annually at 3 anatomical sites (lumbar spine, total hip, and wrist).
  Hypothesis: Relative to women using DMPA only (without tenofovir exposure) and women using PrEP only (without DMPA exposure), women concurrently using TDF-based PrEP and DMPA will have lower bone mass.
The investigators will assess whether young women using TDF-based PrEP and DMPA concurrently have evidence of disrupted microarchitecture, relative to women using either agent singly or neither agent. | 24 months
  The investigators will use dual energy x-ray absorptiometry (DXA) scans to derive the trabecular bone score (TBS), an index of lumbar spine trabecular microarchitecture.
  Hypothesis: Relative to women using DMPA only (without tenofovir exposure) and women using PrEP only (without DMPA exposure), women concurrently using TDF-based PrEP and DMPA will have more disruptions in bone microarchitecture.

SECONDARY OUTCOMES:
The investigators will investigate whether young women concurrently using TDF-based PrEP and DMPA experience higher rates of bone turnover. | Change from Baseline at 24 months
  At baseline and 24 months, the investigators will measure:
  Markers of bone formation and resorption (e.g. NTX, P1NP, serum intact parathyroid hormone, total and bioavailable 25-OH-vitamin D).
  Hypothesis: Relative to women using DMPA only and PrEP only, women concurrently using TDF-based PrEP and DMPA will have increased bone turnover markers and PTH.
The investigators will investigate whether young women concurrently using TDF-based PrEP and DMPA experience higher rates of subclinical kidney injury. | Change from Baseline at 24 months
  At baseline and 24 months, the investigators will measure: Markers of kidney function (phosphate, glucose, creatinine, total protein, albumin).
  Hypothesis: Relative to women using DMPA only and PrEP only, women concurrently using TDF-based PrEP and DMPA will have more frequent subclinical kidney injury (relative to women without tenofovir exposure)
The investigators will investigate whether young women concurrently using TDF-based PrEP and DMPA experience higher rates of hypoestrogenism. | Change from Baseline at 24 months
  At baseline and 24 months, the investigators will measure: Markers of estrogen (serum estradiol, sex hormone binding protein, and the occurrence of amenorrhea).
  Hypothesis: Relative to women using DMPA only and PrEP only, women concurrently using TDF-based PrEP and DMPA will have reduced serum estrogen (relative to women without DMPA exposure).
Using mediation analysis, the investigators will identify the degree to which the pathways through subclinical kidney injury and hypoestrogenism account for changes in bone density among women concurrently using TDF-based PrEP and DMPA | 24 months
  The investigators will conduct mediation analysis to determine the degree to which changes in the pathways through subclinical kidney injury, hypoestrogenism and the combination of these pathways account for changes in bone density.
  Hypothesis: The pathway through hypoestrogenism will be a stronger link between concurrent TDF-based PrEP and DMPA use and bone density changes.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Heffron, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- Infectious Disease Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu L, Ssebuliba T, Muwonge TR, Bambia F, Stein G, Nampewo O, Sapiri O, Goetz BJ, Penrose KJ, Parikh UM, Mujugira A, Heffron R. Alignment of PrEP Use With Potential HIV Exposure in Young Women and Men in Uganda. J Acquir Immune Defic Syndr. 2025 Apr 1;98(4):326-333. doi: 10.1097/QAI.0000000000003573. Epub 2025 Feb 19. PMID 39630076
- [Derived] Zia Y, Nambala L, Stalter RM, Muwonge TR, Ssebuliba T, Nakyanzi A, Nampewo O, Boyer J, Morrison S, Nsubuga R, Bagaya M, Nyanzi R, Matovu F, Yin M, Wyatt C, Mujugira A, Heffron R for the Kampala Women's Bone Study. Depression and PrEP uptake, interruption, and adherence among young women in Uganda. AIDS Care. 2023 Sep;35(9):1365-1374. doi: 10.1080/09540121.2023.2177250. Epub 2023 Mar 9. PMID 36892945

DOCUMENTS (1):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT03464266/Prot_001.pdf